CLINICAL TRIAL: NCT04497272
Title: Assesment of the Metabolomic Signature in COVID-19 Patients (SignCov Study)
Brief Title: Assesment of the Metabolomic Signature in COVID-19 Patients
Acronym: SignCov
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-PP-18
Record Dates: First submitted 2020-08-03; First posted 2020-08-04 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-05

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patient with COVID-19 disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The metabolomic signature of COVID-19 patients (Other): It will consist in the collection of 1 additional tubes at their blood draw and 1 urine sample.
  Interventions: Other: COVID-19 patients

INTERVENTIONS:
Other: COVID-19 patients — It will consist in the collection of 1 additional tubes at their blood draw and 1 urine sample.

SUMMARY:
Metabolomics is the analysis of small molecules in a biological sample (cells, tissues or biological fluids). It can potentially detect very sensitively any change related to a pathology or exposure to a toxic agent. The analyses are fast, inexpensive and therefore applicable in routine, particularly in health care. Given the emergence of this new disease, COVID-19, there is a real need to better understand the pathophysiological mechanisms of SARS-CoV-2 infection. In this context, metabolomics could have a place and could lead to the development of interesting diagnostic or prognostic tools. The objective of this study is to identify, through the analysis of biological samples (blood and urine), whether there is a metabolomic signature in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years of age
* affiliated to a social security scheme
* consultant in the emergency department and/or being hospitalized for suspected SARS CoV infection
* confirmation, after medical examination, of the need for a biological examination (this will negate the need for additional venipuncture)

Exclusion criteria:

* Patient who do not meet inclusion criteria
* Person subject to a guardianship order
* Opposition to the use of the data or samples (withdrawal of non-opposition) / Sponsor's or investigator's decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Identifying the metabolomic signature | Enrollment
  To dentified a metabolomic profile using liquid chromatography combined with mass spectrometry (LC-MS) on the serum and urine of COVID-19 patients

SECONDARY OUTCOMES:
Identification of the metabolomic profile according to clinical severity. | Enrollment
  Identification of the metabolomic profile of patients infected with SARS CoV 2 in the following subgroups: pauci-symptomatic patients, symptomatic patients without clinical severity criteria, and critically ill COVID-19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: OCCELLI Céline, Principal Investigator — Néphrologie, CHU de Nice
Locations (1):
- CHU de nice, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: No